CLINICAL TRIAL: NCT06299124
Title: A Phase I Study Evaluating Safety and Tolerability of RGT-419B Monotherapy in Chinese Patients With Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Advanced/Metastatic Breast Cancer or Other Solid Tumors
Brief Title: A Phase I Study of RGT-419B in Patients With HR-Positive, HER2-Negative Advanced Breast Cancer or Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGT-419B-102
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Bulk Drugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RGT-419B monotherapy (Experimental): Dose escalation and dose expansion of RGT-419B monotherapy
  Interventions: Drug: RGT-419B

INTERVENTIONS:
Drug: RGT-419B — RGT-419B will be administered orally
  Other Names: Active drug

SUMMARY:
This is a Phase 1 dose escalation and dose expansion phase I study to evaluate the safety, tolerability, pharmacokinetic profile and preliminary efficacy of RGT-419B as monotherapy in Chinese patients with HR+/HER2- advanced/metastatic breast cancer and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Subjects with pathologically confirmed advanced solid tumors who have failed standard-of-care therapy, or have no standard-of-care therapy available, or are currently not eligible for standard-of-care therapy; Subjects with HR+/ HER2- advanced or metastatic breast cancer are preferred.
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Presence of visceral metastases with severe organ dysfunction
* Known active hepatitis B or C infection
* Prior irradiation to >25% of the bone marrow and/or inadequate bone marrow function or evidence of clinicallysignificant end-organ damage
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs usedin the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety & Tolerability - Number of subjects with Dose-Limiting Toxicities (DLTs) at each cohort dose level | 4 weeks (1 cycle)
  Number of subjects who have a confirmed DLT at each cohort dose level during the first 28-day cycle of RGT-419B treatment.

SECONDARY OUTCOMES:
Safety & Tolerability - Incidence, Severity, and Causality of all Treatment Emergent Adverse Events (TEAEs) | through study completion, an average of 1 year
  Incidence, severity, and causality of all TEAEs will be assessed for all patients participating from Day 1 dosing through end of study.
Day 1 and steady-state pharmacokinetics(PK) assessment of RGT-419B and major metabolites - Cmax | 4 weeks (1 cycle)
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Area Under Concentration-TimeCurve to Infinity (AUC0-inf) | 4 weeks (1 cycle)
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Plasma Decay Half-Life (t1/2) | 4 weeks (1 cycle)
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Time to Reach Maximum ObservedPlasma Concentration (Tmax) | 4 weeks (1 cycle)
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Accumulation rate after multipledoses | 4 weeks (1 cycle)
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Cumulative urinary excretion | 4 weeks (1 cycle)
Tumor Response assessed by Investigator according to RECIST v1.1 | through study completion, an average of 1 year
QTc Interval - Changes in corrected QT interval | through study completion, an average of 1 year
  Number of subjects with a clinically significant increase from baseline in corrected QT (QTc) interval onrepeated ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No